CLINICAL TRIAL: NCT05415813
Title: Effects of Ischemic Compression With and Without Muscle Energy Technique on Pain, Range of Motion and Functional Disability in Patients With Trigger Points in Upper Trapezius; A Randomized Clinical Trial
Brief Title: Effects of IC With and Without MET on Upper Trapezius Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/890-II/2021
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Upper Trapezius Trigger Points
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Compression (Active Comparator): Ischemic Compression will be applied to the upper trapezius trigger points in patients recruited in group 1.
  Interventions: Other: Ischemic Compression
- Ischemic compression and Muscle Energy Technique (Experimental): ischemic compression along with muscle energy technique will be applied to the upper trapezius trigger points in patients allocated to group 2.
  Interventions: Other: Ischemic compression with Muscle Energy Technique

INTERVENTIONS:
Other: Ischemic Compression — It includes conventional Physical therapy, hot packs (75°C) for 20 minutes, and active stretching exercises for the upper trapezius muscle (slow, 5 repetitions per session, 10-second hold, and 10-second relaxation between two repetitions) as a baseline treatment. For the Ischemic compression, the patient will be in the supine position with the cervical spine in opposite lateral flexion to the treating part so that the upper trapezius muscle fibers were kept in a lengthened position physiotherapist will apply gradually increasing pressure to the Trigger points until the subject perceived the first noticeable pain. At that moment, the pressure will be maintained until the discomfort and/or pain eased by around 50% as perceived by the patient, at which time the pressure will be increased until the discomfort appears again. This process will be maintained for 90 seconds.
  Arms: Ischemic Compression
Other: Ischemic compression with Muscle Energy Technique — The Participants will receive all the treatments given to the active comparator group and they will also receive the Muscle Energy Technique treatment in supine position and the practitioner will stabilize the shoulder of the affected side with one hand, while the ear/mastoid area of the affected side will be held by the opposite hand. The head and neck were then bent towards the contralateral side, flexed, and ipsilaterally rotated. The subjects will then shrug the stabilized shoulder towards the ear at a sub-maximal pain-free effort (20% of the available strength). The isometric contraction will be held for 7-10s. This position will be maintained for 30 seconds and repeated three to five times per treatment session. Treatment sessions will be given on alternate days.
  Arms: Ischemic compression and Muscle Energy Technique

SUMMARY:
the aim of the study is to check the effects of ischemic compression with and without muscle energy technique on Pain, Range of motion, and Functional Disability on myofascial trigger points in the upper trapezius. In previous studies, Muscle Energy Technique and Ischemic Compression are compared with different conventional and combined therapy approaches, including most of the techniques used to treat Trigger Points in the upper trapezius. No study has evaluated the effects of ischemic compression with and without muscle energy technique on Pain, Range of motion, and Functional Disability on myofascial trigger points in the upper trapezius. The outcome measures are a Numeric pain rating scale, universal goniometer and neck disability index questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Both gender Aged 18 to 50 years (40)
* Participants with active myofascial trigger points in the upper trapezius diagnosed by a senior physiotherapist on the basis of Travel and Simon criteria will be randomly allocated into two clinical groups.
* Taut band having palpable nodule within upper trapezius muscle
* Pain produced in a specific pattern which is radiating in character when firm pressure is applied on trigger points

Exclusion Criteria:

* Trauma (whiplash injury)
* Injury to Cervical Spine
* Cervical Spine surgery
* Cervical Myelopathy and Radiculopathy
* Osteoporosis of the cervical spine
* Cervical myeloma
* Complex regional pain syndrome
* Patients with the H/O any Neurological, Rheumatology and other serious medical illnesses.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in pain on Numeric Pain Rating Scale at week 4 | Baseline and week 4
  on a scale of 1 to 10, o means no pain while 10 means worst pain
Change from Baseline in Goniometer readings at week 4 | Baseline and week 4
  for flexion any value less than 90 degrees indicates limited range of motion, for extension any value less than 70 indicates limited range of motion, for lateral flexion values less than 20 and greater than 45 considered limited, for rotation value less than 90 is considered limited
Change from baseline in Neck disability index questionnaire scores at week 4 | Baseline and week 4
  on a scale of 0 to 50, 0 indicates no disability and 50 indicates completely disabled

SECONDARY OUTCOMES:
Pain on Numeric Pain Rating Scale at week 2 | week 2
  on a scale of 1 to 10, o means no pain while 10 means worst pain
Goniometer readings at week 2 | week 2
  Using goniometer, neck ranges of motion will be measured. for flexion any value less than 90 degrees indicates limited range of motion, for extension any value less than 70 indicates limited range of motion, for lateral flexion values less than 20 and greater than 45 considered limited, for rotation value less than 90 is considered limited
Neck disability index questionnaire scores at week 2 | week 2
  on a scale of 0 to 50, 0 indicates no disability and 50 indicates completely disabled

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Khadija Kazmi, DPT, Principal Investigator — University of Lahore
Locations (1):
- University of Sialkot, Sialkot, Punjab Province, Pakistan